CLINICAL TRIAL: NCT07076316
Title: Effects of a Structured Early Rehabilitation Nursing Pathway on Gastrointestinal Recovery and Quality of Life in Severe Acute Pancreatitis Patients: A Randomized Controlled Trial
Brief Title: Early Rehabilitation Nursing for Severe Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qiandi Huang (Other)
Responsible Party: Sponsor-Investigator, Qiandi Huang, Principal investigator, Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University
Organization: Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHUSH-SAP-ERN-2021-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Pancreatitis Drug-Induced
Keywords: Early Rehabilitation Nursing; Severe Acute Pancreatitis; Patient-Centered Care; Functional Recovery; Critical Care; Quality of Life
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERN Group (Experimental): Patients received a structured early rehabilitation nursing pathway (SERNP) in addition to routine care. The intervention was implemented within 48 hours of hemodynamic stability and included:
  * Phase 1 (Days 1-3): Bedside passive range-of-motion exercises (10 min/session, 2x/day), respiratory training (lip pursing and abdominal breathing, 3 sessions/day), and gradual head-of-bed elevation (30° to 90°).
  * Phase 2 (Days 4-7): Progressive mobilization including sitting at bedside (5-10 min, 3x/day) and assisted standing with a tilt-table (≤15 min/session).
  * Phase 3 (Days 8-14): Supervised ambulation (2-5 meters, 2x/day) with mobility aids.
  Interventions: Behavioral: Structured Early Rehabilitation Nursing Pathway
- Control Group (Active Comparator): Patients received routine care, which included vital sign monitoring, strict fasting, fluid balance recording, and passive limb mobilization twice daily.
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Structured Early Rehabilitation Nursing Pathway — A multi-component, phased nursing intervention focused on early and progressive mobilization, respiratory exercises, and psychological support.
  Arms: ERN Group
Behavioral: Routine Care — Standard nursing care for severe acute pancreatitis patients in the ICU, including monitoring and passive limb mobilization.
  Arms: Control Group

SUMMARY:
This randomized controlled trial evaluates the clinical efficacy of a structured early rehabilitation nursing (ERN) pathway compared to routine care in patients with severe acute pancreatitis (SAP). The study aims to determine if the ERN pathway, which includes phased mobility, respiratory training, and psychological support, can improve gastrointestinal recovery, reduce hospital stay and complications, and enhance functional independence and quality of life.

DETAILED DESCRIPTION:
Severe acute pancreatitis (SAP) is a life-threatening condition with high mortality and morbidity, often complicated by prolonged immobilization, leading to muscle atrophy, delayed gut recovery, and increased infection risk. Current nursing practices often neglect early mobilization. This study introduced and tested a structured early rehabilitation nursing pathway (SERNP) designed to address these gaps. A total of 104 eligible SAP patients were randomly assigned to either the SERNP group (n=52) or a control group receiving routine care (n=52). The SERNP intervention was initiated within 48 hours of achieving hemodynamic stability and was delivered in three phases over 14 days: Phase 1 (Days 1-3) focused on bedside passive exercises and respiratory training; Phase 2 (Days 4-7) introduced progressive mobilization like sitting and assisted standing; and Phase 3 (Days 8-14) involved supervised ambulation. The study hypothesis was that the SERNP would accelerate recovery and improve outcomes by addressing both the physiological and psychosocial consequences of SAP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Severe Acute Pancreatitis (SAP) according to the Revised Atlanta Classification.
* APACHE II score > 8.
* Expected ICU stay ≥ 14 days.
* Hemodynamic stability (mean arterial pressure ≥ 65 mmHg for > 24 hours).
* Provided informed consent.

Exclusion Criteria:

* Presence of chronic metabolic disorders (e.g., end-stage renal disease, cirrhosis).
* Coagulopathy (INR > 1.5 or platelet count < 50×10⁹/L).
* Cognitive impairment hindering cooperation with the rehabilitation protocol.
* Recent use of antiplatelet or anticoagulant medication (within 7 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Time to Relief of Abdominal Distension | From randomization up to hospital discharge (an average of 14 days)
  Time in days from randomization until the resolution of abdominal distension, as assessed by clinical evaluation.
Time to First Bowel Movement | From randomization up to hospital discharge (an average of 14 days)
  Time in days from randomization until the first anal exhaust (bowel movement).
Duration of Hospital Stay | From hospital admission up to hospital discharge (an average of 14 days)
  Total length of stay in the hospital, measured in days.
Incidence of Complications | From randomization until hospital discharge (an average of 14 days)
  Percentage of patients who developed complications, including pressure ulcers, pneumonia, and venous thrombosis.

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) Score | Within 24 hours prior to Intensive Care Unit (ICU) discharge
  Functional independence measured using the Barthel Index (BI). The scale ranges from 0 to 100, with higher scores indicating greater independence.
Quality of Life (QoL) Score | At 48 hours prior to hospital discharge
  Quality of life assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire. This measures four domains: physical health, psychological health, social relationships, and environment. Scores are transformed to a 0-100 scale, with higher scores indicating better QoL.
Nursing Satisfaction | Within 24 hours prior to hospital discharge
  Patient satisfaction with nursing care, measured using a 10-item Likert scale developed for ICU settings. The rate of patients rating care as "satisfied" or "very satisfied" was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jianghan University, The Sixth Hospital of Wuhan, Wuhan, Hubei, China